CLINICAL TRIAL: NCT05500339
Title: CARE 1000. Randomized Control Trial for the Evaluation of the Effectiveness of a mHealth App for Supporting the First 1000 Days of Life
Brief Title: Effectiveness of a mHealth App for Supporting the First 1000 Days of Life
Acronym: CARE1000
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC 04\2022
Record Dates: First submitted 2022-08-04; First posted 2022-08-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Health-Related Behavior
Keywords: mHealth application; first 1000 days; health prevention
MeSH Terms: conditions — Health Behavior | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth App (Experimental): The mHealth App designed for the support of the first 1000 days of life is provided to pregnant women. Specific contents are presented to the user according to the current trimester of pregnancy or the post-partum period following a scheduled routine; all contents are always available for free consultation during the entire period of use. Links to relevant institutional websites are also reported for any further reading. The app has a frequently asked question (FAQ) section, and a calendar function with the possibility to set appointments and reminders. App contents and topics include information about health prevention behaviors such as vaccination during pregnancy, weight increment during pregnancy, abstinence from smoke and alcohol consumption habits, adherence to child routine vaccination schedule.
  Interventions: Other: M-health App
- Standard care. (Sham Comparator): Pregnant women receive standard supportive and educational methods.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: M-health App — Pregnant women receive the App designed for the support of the first 1000 days of life
  Arms: mHealth App
Other: Standard care — Pregnant women receive standard supportive and educational methods.
  Arms: Standard care.

SUMMARY:
Recent development in information and communication technologies has enabled the disruptive expansion of electronic health (eHealth) and mobile health (mHealth). These developments, along with the introduction in clinical practice of technological innovations, such as telemedicine, telemonitoring, and remote screening, are considered essential elements of "game-changing innovations" in the next 25 years. In fact, the widespread distribution of networked devices, which are estimated to reach 29.3 billion in 2023, offers a promising but challenging opportunity of mHealth use for health information seeking, with an important role in health behavior formation. In 2017, more than 325,000 mobile health applications (apps) were available worldwide, and among them, to the best of our knowledge, there were more apps available to support pregnancy than for any other medical domain. These mobile technologies in support of pregnancy have also increased the possibility for both parents and parents-to-be to self-manage health issues; findings from a recent study conducted in 2019 in Switzerland report that 91% of parents declared using digital media for seeking information about their child's health and development. Moreover, a recent meta-analysis showed that social media and mHealth have the potential to be effective in promoting maternal physical health (e.g., weight management), mental health, and knowledge about pregnancy. However, when considering apps addressing children's first 1000 days of life, from conception through age 24 months, many of them just focus on the prenatal or postnatal stage, failing to consider the continuity between the two phases and their joint impact on maternal and child health.

The purpose of this study is to evaluate the mHealth App effectiveness for the support of women during the first 1000 days (from conception through age 24 months) and for improving health prevention behaviors such as vaccination during pregnancy, weight increment during pregnancy, abstinence from smoke and alcohol consumption habits, adherence to child routine vaccination schedule.

In addition, the study aims to understand the level of appreciation of this mHealth App as a tool to overcome information and communication gaps between patients and institution.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women accessing for the first trimester ultrasound.
* Age >= 18 years
* Good comprehension of Italian language
* Possession of a smartphone for the App download
* Willingness to give birth at Institute for Maternal and Child Health Burlo Garofolo, Trieste

Exclusion Criteria:

- Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Between groups differences in the adherence of pregnant women to Tetanus, Diphtheria, Pertussis (TDaP) vaccination | Within the second year of child life
  Number of vaccination in pregnancy carried out in the two groups

SECONDARY OUTCOMES:
Between groups differences in women knowledge | Immediately at the end of first trimester of pregnancy
  Differences between experimental and control group in health prevention and promotion knowledge evaluated with questionnaire (closed questions with the following possibile answers: true/false/I don't know)
Between groups differences in women behaviors | Immediately at the end of first trimester of pregnancy
  Differences between experimental and control group in health prevention and promotion behaviors evaluated with questionnaire (questions with five-level Likert scale answers from 1 to 5, when 1=Strongly disagree and 5=Strongly agree)
Between groups differences in women knowledge | At the end of second trimester of pregnancy
  Differences between experimental and control group in health prevention and promotion knowledge evaluated with questionnaire (closed questions with the following possibile answers: true/false/I don't know)
Between groups differences in women behaviors | At the end of second trimester of pregnancy
  Differences between experimental and control group in health prevention and promotion behaviors evaluated with questionnaire (questions with five-level Likert scale answers from 1 to 5, when 1=Strongly disagree and 5=Strongly agree)
Between groups differences in women knowledge | Within the second year of child life
  Differences between experimental and control group in health prevention and promotion knowledge evaluated with questionnaire (closed questions with the following possibile answers: true/false/I don't know)
Between groups differences in women behaviors | Within the second year of child life
  Differences between experimental and control group in health prevention and promotion behaviors evaluated with questionnaire (questions with five-level Likert scale answers from 1 to 5, when 1=Strongly disagree and 5=Strongly agree)
Between groups differences in Health literacy level | Immediately at the end of first trimester of pregnancy
  Differences between experimental and control group in Health literacy level measured with the Italian version of the 16-items European Health Literacy Survey Questionnaire (HLS-EU-Q16)
Between groups differences in Health literacy level | Immediately at the end of second trimester of pregnancy
  Differences between experimental and control group in Health literacy level measured with the Italian version of the 16-items European Health Literacy Survey Questionnaire (HLS-EU-Q16)
Between groups differences in Health literacy level | Within the second year of child life
  Differences between experimental and control group in Health literacy level measured with the Italian version of the 16-items European Health Literacy Survey Questionnaire (HLS-EU-Q16)
Between groups differences in social and health impact | Within the second year of child life
  Differences between experimental and control group in social and health impact evaluated with questionnaire (i.e., number and type of contacts with health services; time spent on internet to collect health information and ease of information retrieval; ease of sharing information on pregnancy and post-partum within the household; ability to manage health during pregnancy and in the post-partum period)
Appreciation of the mHealth App | Within the second year of child life
  Only for the experimental group, appreciation of the mHealth app to bridge the information gap between citizens and health institutions, evaluated with questionnaire
MHealth app usage data | Within the second year of child life
  Collection of data about App usage for the experimental group, i.e., App access frequency, content consultation, references consultation, App features use

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Stampalija, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

REFERENCES:
- [Derived] Brunelli L, Bussolaro S, Dal Cin M, Ronfani L, Zanchiello S, Cassone A, Verardi G, Dobrina R, Bava M, Stampalija T. CARE 1000: randomized controlled trial for the evaluation of the effectiveness of a mHealth app for supporting the first 1000 days of life. Trials. 2022 Dec 12;23(1):1007. doi: 10.1186/s13063-022-06953-y. PMID 36510286